CLINICAL TRIAL: NCT02765724
Title: A Phase 1 Open Label, Single Dose, Parallel-Group Study to Determine the Pharmacokinetics of Pacritinib in Patients With Impaired Hepatic Function in Comparison With Healthy Subjects
Brief Title: Determine Pacritinib Pharmacokinetics in Impaired Hepatic Patients and Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CTI BioPharma (Industry)
Collaborators: SGS S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PAC103
Record Dates: First submitted 2016-05-03; First posted 2016-05-09 (Estimated); Last update posted 2020-03-06 (Actual); Status verified 2016-05

CONDITIONS: Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene

ARMS (4):
- Group 1 (Experimental): Patients with mild hepatic impairment
  Interventions: Drug: Pacritinib
- Group 2 (Experimental): Patients with moderate hepatic impairment
  Interventions: Drug: Pacritinib
- Group 3 (Experimental): Patients with severe hepatic impairment
  Interventions: Drug: Pacritinib
- Group 4 (Experimental): Healthy subjects
  Interventions: Drug: Pacritinib

INTERVENTIONS:
Drug: Pacritinib — Pacritinib 400 mg (4 capsules of 100 mg each), single dose, oral administration
  Other Names: Pacritinib 400mg capsule

SUMMARY:
This is an open-label, parallel-group, single-dose study of the PK and safety of 400 mg pacritinib administered orally to patients with stable chronic liver disease and healthy control subjects.

DETAILED DESCRIPTION:
All study participants will undergo screening evaluations to determine eligibility for the study. All screening evaluations must be performed within 28 days of pacritinib dosing (Day 1). Assignment of patients to each hepatic impairment group will be defined by Child-Pugh Clinical Assessment Score at the time of Screening. Group 3 patients will not be dosed until at least 2 patients combined from Groups 1 and 2 have completed the study (Day 8). Healthy subjects will be enrolled after hepatic impairment accrual is complete to allow for age-, gender- and body mass index- (BMI) matching with the hepatic impairment population. Participants will be admitted to the study site on Day -1 (i.e., Check-in). On Day 1, upon receipt of all baseline safety evaluation results and confirmation of eligibility, study participants will be administered a single dose of 400 mg pacritinib orally under fasting conditions. Fasting will start 10 hours prior to pacritinib administration and continue for an additional 4 hours after administration. Following administration of pacritinib, participants will remain confined to the study site for 168 hours (8 days) after pacritinib dosing for collection of blood for PK and safety assessments.

ELIGIBILITY:
Inclusion Criteria:

All Study Participants

1. Male and/or female from 18-85 years of age, inclusive
2. Must be in sufficiently good health to tolerate the study treatment and procedures and be evaluable for possible effects of hepatic dysfunction on pacritinib PK without significant confounding issues, in the opinion of the investigator in consultation with the Sponsor
3. Must be using a medically-approved birth control method

   * Females must be non-pregnant and non-lactating, and females not of childbearing potential must be postmenopausal for at least 1 year or surgically sterile (e.g., tubal ligation, hysterectomy) for at least 90 days, or agree to use, from the time of signing the informed consent or 10 days prior to Check-in (Day -1) until 30 days after Study Completion (Day 8)/Early Termination, one of the following forms of contraception: non-hormonal intrauterine device (IUD) with spermicide; female condom with spermicide; contraceptive sponge with spermicide; intravaginal system (e.g., NuvaRing®); diaphragm with spermicide; cervical cap with spermicide; male sexual partner who agrees to use a male condom with spermicide; sterile sexual partner; or abstinence. Oral, implantable, transdermal, or injectable contraceptives may not be used from the time of signing the informed consent or 10 days prior to Check-in (Day -1) until 14 days after the final dose administration. For all females, the pregnancy test result must be negative at Screening and Check-in (Day -1)
   * Males will be sterile, or completely abstain from sexual intercourse, or agree to use, from Check-in (Day -1) until 90 days following Study Completion/ET, one of the following approved methods of contraception: male condom with spermicide; sterile sexual partner; or use by female sexual partner of an IUD with spermicide; a female condom with spermicide; a contraceptive sponge with spermicide; an intravaginal system; a diaphragm with spermicide; a cervical cap with spermicide; or oral, implantable, transdermal, or injectable contraceptives. Study participants will refrain from sperm donation from Check-in (Day -1) until 90 days following Study Completion (Day 8)
4. BMI between 18-40 kg/m2 (inclusive) at Screening
5. Vital signs (after 3 minutes seated position rest then measured in the seated position) within the following ranges, inclusive, unless deemed not clinically significant by the Investigator, as approved by the Sponsor:

   * oral body temperature between 35.0-37.5 °C
   * systolic blood pressure, 90-160 mm Hg
   * diastolic blood pressure, 50-100 mm Hg
   * pulse rate, 50-100 bpm

   Blood pressure and pulse will be taken again in a standing position. After 3 minutes standing, there shall be no more than a 20 mm Hg drop in systolic blood pressure associated with symptomatic postural hypotension
6. Negative test for selected drugs of abuse (including alcohol) at Screening and at Baseline, prior to admission to study site, except for positive tests due to prescribed drugs in hepatic impaired patients
7. Negative human immunodeficiency virus (HIV) antibody screens
8. Able to communicate well with the investigator, to understand and comply with the requirements of the study. Understand and sign the written informed consent. Legal authorized representatives are not permitted

   Patients with Hepatic Impairment Only
9. Child-Pugh Clinical Assessment Score consistent with degree of hepatic impairment that is not attributable to any other underlying disease
10. Patients assigned to a hepatic impairment group must be evaluable and meet criteria for hepatic impairment per the Child-Pugh Clinical Assessment Score

    Healthy subjects only
11. Healthy subjects will be identified after all hepatic impairment patients have been enrolled and the healthy subject group will have similar distributions of age (by hepatic impairment population quartiles), BMI (by hepatic impairment population quartiles) and gender
12. Negative hepatitis panel (including hepatitis B surface antigen [HBsAg], hepatitis B core antibody (anti-HBc), and hepatitis C virus antibody [anti-HCV])

Exclusion Criteria:

Study participants meeting any of the following criteria during Screening or Baseline evaluations will be excluded from entry into or continuation in the study:

All Study Participants

1. Participation in any clinical investigation within 4 weeks prior to Check-in or longer if required by local regulation
2. Participation in any clinical investigation involving receipt of investigational study drug within 5 half-lives or 30 days prior to Check-in (Day -1) (whichever is longer)
3. Donation or loss of 400 mL or more of blood within 8 weeks prior to Check-in
4. Significant illness within the two weeks prior to Check-in
5. A past medical history of clinically significant ECG abnormalities, presence of an abnormal ECG (which in the Investigator's opinion is clinically significant), QTcF >450 msec, or has concomitant conditions that significantly increase risk for QTc interval prolongation such as heart failure or family history of long QT interval syndrome)
6. Resting heart rate < 50 beats per minute (bpm)
7. Alcohol ingestion within 72 hours of Check-in
8. Urine Cotinine levels ≥ 150 ng/mL
9. Use of potent inducers of CYP3A4 (Appendix 4) within 30 days of Check-in
10. Use of potent inhibitors of CYP3A4 (Appendix 4) within 15 days of Check-in
11. Use of over-the-counter medications (except as prescribed by a physician), vitamins, or phytotherapeutic/herbal/plant-derived preparations within 14 days of Check-in
12. Consumption of grapefruit- and grapefruit-containing products is not permitted within 7 days of Check-in
13. History of clinically significant drug allergy; history of atopic allergy (asthma, urticaria, eczematous dermatitis). A known hypersensitivity to the study drug, study drug excipients, or drugs similar to the study drug
14. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs or which may jeopardize the study participant in case of participation in the study. The investigator should be guided by evidence of any of the following:

    * history of inflammatory bowel syndrome
    * recent history (within 1 year) of ongoing gastritis or ulcers
    * history of major gastrointestinal tract surgery such as gastrectomy, gastroentero- stomy, or bowel resection (esophageal varix surgery is allowable)
    * clinical evidence of pancreatic injury or pancreatitis
    * evidence of urinary obstruction or difficulty in voiding at Screening
15. History of immunocompromise, including a positive HIV test result

    Patients with Hepatic Impairment Only
16. Clinically significant abnormal findings in physical examination, ECG or laboratory evaluations not consistent with known clinical disease
17. Symptoms or history of Stage II or worse degree of encephalopathy within 6 months of study entry as judged by the investigator
18. Clinical evidence of severe ascites: ascites causing marked abdominal distension and/or being refractory to medical therapy
19. History of surgical portosystemic shunt
20. Neutrophil count <1500/mm3, Platelet count <30,000/mm3, Hemoglobin <9 g/dL
21. Prothrombin time > 18 seconds
22. Creatinine clearance (CrCl) of less than 60 ml/min as calculated by the Cockcroft-Gault equation ((140-age in years) × (Weight in kg) × (0.85 if female) / (72 × Serum Creatinine in mg/dL))
23. Any evidence of progressive liver disease (as available within the last 4 weeks, including the time period between Screening and Check-in) as indicated by liver transaminases, alkaline phosphatase, and gamma-glutamyl transpeptidase or a ≥ 50% worsening of serum bilirubin or prothrombin time
24. Urinalysis with any result outside the normal range and deemed clinically significant. Results deemed not clinically significant by investigator in consultation with the Sponsor are allowable
25. Initiation of any otherwise allowable prescription or over-the-counter medications within 15 days of Check-in. Some of these medications may have to be discontinued 12 to 48 hours pre-dose, or earlier. As medication regimens vary and cannot be predicted, each patient shall be discussed with the Sponsor individually
26. History of drug or alcohol abuse within the last 3 months, or evidence of recent drug or alcohol abuse in alcohol test and drug screen conducted during Screening or Baseline evaluations

    Healthy Subjects Only
27. Any Screening or Baseline laboratories outside the normal range and deemed clinically significant. Results outside the normal range and deemed not clinically significant by investigator, in consultation with the Sponsor, are allowable
28. History of drug or alcohol abuse within the last 12 months, or evidence of such abuse as indicated by the laboratory assays conducted during the Screening or Baseline evaluations
29. Use of any prescription medication within 1 month prior to Check-in

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
To characterize the pharmacokinetic profile of a single 400-mg dose of pacritinib and its major metabolites in patients with hepatic impairment as compared to gender-, age-, and body mass index -matched healthy subjects with normal liver function | Plasma: 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose
  Plasma concentrations of pacritinib and any major metabolites were determined by a validated, sensitive, and specific high performance liquid chromatography/tandem mass spectrometric assay. The lower limit of quantitation of the assay is 20 ng/mL for pacritinib and 4 ng/mL for PAC-M1 metabolite in plasma

SECONDARY OUTCOMES:
To evaluate the safety of pacritinib and tolerability of a single 400-mg dose of pacritinib in patients with hepatic impairment and healthy subjects; | 00:00 of ICF signature until 1 min before IP admin and from the date-time of IP administration until 23:59 of the day of last contact
  Adverse events, vital signs, physical examinations, clinical laboratory valuations, and ECGs

CONTACTS AND LOCATIONS:
Overall Officials: James Dean, MD, PhD, Study Director — CTI BioPharma
Locations (2):
- APEX GmbH, Munich, Germany
- Republican Clinical Hospital, Chisinau, Moldova

IPD SHARING:
Plan to Share IPD: Yes